CLINICAL TRIAL: NCT03911180
Title: Pertrochanteric Fracture Fixation In Elderly Adults Using Proximal Femoral Nail Anti-rotation (HERACLES) With a T-shaped Parallel Blade: A New Design
Acronym: Heracles PFN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ilocos Training and Regional Medical Center (Other Government)
Responsible Party: Principal Investigator, Lou Mervyn Tec, Orthopedic Resident Year Level IV, Ilocos Training and Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITRMCOrthoCS0001
Record Dates: First submitted 2019-04-06; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Pertrochanteric Fracture; Intertrochanteric Fractures; Pertrochanteric Fracture of Femur, Closed; Pertrochanteric Fracture of Femur, Open
Keywords: Pertrochanteric fracture; Intertrochanteric fracture; subtrochanteric extension; Proximal femoral nail; Proximal locking screw; Distal locking screw
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PFN straight parallel blade (Experimental): All patients with pertrochanteric fracture that is eligible will undergo PFNA with straight parallel blade.
  Interventions: Device: Proximal femoral nail with straight parallel blade

INTERVENTIONS:
Device: Proximal femoral nail with straight parallel blade — Petrochanteric fixation with Heracles proximal femoral nail
  Other Names: Heracles proximal femoral nail

SUMMARY:
This is a prospective case series of elderly adult patients sustaining pertrochanteric fractures who will be treated by a proximal femoral nail with a non-helical (straight) blade. This study seeks to observe and evaluate the outcomes, advantages and complication rates in using the HERACLES PFN with a non-helical (T-shaped parallel) blade.

DETAILED DESCRIPTION:
The trochanteric area is defined by AO as the area bordered by the tip of the greater trochanter, extracapsular portion of the femoral neck extending to a line parallel to the inferior most border of the lesser trochanter.

Pertrochanteric fracture is a fracture is of the trochanteric area which is usually reducible. Unstable pertrochanteric fracture is defined as AO-31A2 or AO-31A3. Instability arises from the degree of comminution, the presence, and comminution of the posteromedial fragment and lastly, lateral wall involvement The ideal implant for fixation of this kind of fractures is still under debate, but intramedullary implants are preferred than extramedullary implants in these unstable fractures. On the other hand, unique fracture configurations predispose to instability such as reverse obliquity fractures and fractures extending to the subtrochanteric area.

Proximal femoral locking plate as used in unstable pertrochanteric fracture has a high complication rate. In one study in 2014, there is up to 41.4% failure rate due to the proud plate, screw malposition, too rigid construct when used as a bridge plate.

Intramedullary implants specifically cephalomedullary nails has been the mainstay of treatment in unstable pertrochanteric fractures primarily because of the short moment arm and load-sharing properties. It employs relative stability and can be applied in a minimally invasive manner.

In 1997, the AO/ASIF group developed the proximal femoral nail. The proximal femoral nail has two proximal screws that traverse the neck to the femoral head. The inferior screw is the load-bearing screw, and the superior screw is the anti-rotation screw. Good to excellent results were observed using this implant compared to previous implant designs, but complications still exist.

These complications are related to the position of the two screws. There is difficulty attaining the ideal placement of proximal locking screws. As a result, the early medial cutout of one screw and lateral migration of the second screw occurs which is the so-called Z-effect. To address these disadvantages, the AO/ASIF group in 2004 developed a new implant design wherein the two proximal locking screws are replaced by a single helical blade. This improvement in design maximizes bone purchase and bone contact in cancellous bone hereby improving cutout rates.

Even with the new PFNA implant is not exempted from complications. Zhou and Chang in 2012 identified 12 cases of helical blade protrusion in 6 papers. Biomechanically, the helical blade migrates axially through the porotic bone in the geriatric population.

The new design of the blade includes a T-shaped anchor for stable fixation in osteoporotic bone. The nail also features a flat lateral design with a smooth radius transition from proximal to distal portion of the nail compared to the bulky profile of conventional nail resulting in easier insertion. Locking mechanism inherent to the nail and blade limits gliding and rotation of the blade. One of the advantages of the system is the use of a radiolucent arm with targeting options for an anti-rotation pin and determination of the superior most aspect of the femoral head for reference.

This case-series introduces a modification in implant design of the PFNA and aims to observe outcomes, advantages, and complications related to its use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sustained stable pertrochanteric fracture (AO31A.1)
2. Patients who sustained unstable pertrochanteric fracture (AO31A.2 or AO31A.)

Exclusion Criteria:

1. Patients who are bedridden
2. Patients with a neurologic/psychiatric disorder (previous or present)
3. Patients with severe dementia/Alzheimer's disease
4. Patient with a history of hip dislocation (whether reduced or unreduced)
5. Patient who underwent previous operation on the hip
6. Patient with amputation of one or both legs
7. Patient with segmental fractures involving the ipsilateral femoral shaft/metaphysis
8. Patient with pathologic fractures, e.g. secondary to metastatic bone disease/ metabolic bone disease
9. Patient presenting with an infection
10. Patient who sustained multiple injuries from other body systems

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical Union | 2 months to 4 months
  Weeks until Union
  Clinical Union - fracture site becomes stable and pain-free
Time to full weightbearing | 4-6 months
  weeks until full weight bearing without pain

SECONDARY OUTCOMES:
Quality and Maintenance of Reduction | up to 2 years
  Acceptable reduction was defined as:
  1. Range of neck angle between 5° varus and 20° valgus.
  2. <20 deg angulation on lateral
  3. No fragment greater than 4 mm displaced
  Reduction is defined as good (3/3), adequate (2/3) and poor (0-1/3)
Tip-Apex Distance | up to 2 years
  expressed in millimetres, is the sum of the distance from the tip of the blade to the apex of the femoral head on both AP and lateral radiographic views
Blood Loss | Taken immediately postop
  Blood loss during the procedure in milliliters
Fluoroscopy time | Intraoperative measurement
  Total time of exposure during the procedure starting from identification of starting point to insertion of distal locking screw
Mobility scale | up to 2 years
  Mobility scoring modified for use in patients who sustained a hip fracture (Bowers and Parker 2016). 1 is best and 10 is worst.
  1. Never uses any walking aid, no restriction in walking distance
  2. Never uses any walking aid, can walk less than one kilometer
  3. Occasionally uses a walking aid
  4. Normally uses one walking stick or needs to hold on to furniture
  5. Normally uses two sticks or crutches
  6. Mobilizes with a frame alone, without the need for assistance
  7. Mobilizes with a frame and the assistance of one other person
  8. Mobilizes with a frame and the assistance of two people
  9. Bed-to-chair, or wheelchair-bound
  10. Bedbound most or all of the day.
Social dependence scale | up to 2 years
  Modified to apply for hip fractures; includes determination of independence to ADLs and advanced ADLs (Bowers and Parker 2016) 1 is best and 8 is worst
  1. Completely independent
  2. Minimal assistance
  3. Moderate assistance
  4. Regular assistance
  5. Dependent
  6. Severely dependent
  7. Fully dependent
  8. Patient temporarily resident in hospital
Pain scale | Postop up to 2 years
  Pain scale adapted for hip fractures (Bowers and Parker 2016) 1 is best and 8 is worst
  0. Unable to answer
  1. No pain at all in the hip
  2. Occasional and slight pain
  3. Some pain when starting to walk, no rest pain.
  4. None or minimal pain at rest, some pain with activities
  5. Regular pain with activities which limits walking distance.
  6. Frequent rest pain and pain at night. Pain on walking.
  7. Constant pain presents around the hip.
  8. Constant and severe pain in the hip requires regular strong analgesia such as opiates.
Radiographic Union Score for the Hip | up to 2 years
  is a validated outcome instrument designed to improve intra and interobserver reliability when describing the radiographic healing of proximal femur fractures
  Based on grading of the anterior cortex, posterior cortex, lateral cortex and medial cortex bridging
  1. - No cortical bridging
  2. - Some cortical bridging
  3. - Complete Cortical Bridging
  In addition, disappearance of the fracture line in the anterior cortex, posterior cortex, medial cortex, lateral cortex
  1. - Fully visible fracture line
  2. - Some evidence of the fracture line
  3. - No evidence of fracture line
  Add all component scores to get the total score
Radiation load | Intraoperative measurement
  Amount of radiation during the procedure as measured by a Dosimeter

OTHER OUTCOMES:
Complications | Intraoperative to postoperative up to 2 years
  Intraoperative and Postoperative complications. Will describe presence of complications and description of the specific complications.
  Intraoperative complications involve redisplacement, iatrogenic fracture and comminution, broken implants (drill bit); These include Infection (superficial or deep); Osteomyelitis; Nonunion; Implant failure; Varus collapse and Others
  Complications will be described in detail to ascertain its causality and recommend how it could have been prevented.
Technical difficulties | Intraoperative
  Technical difficulties encountered during each component step of the OR These include difficulty in finding the entry point; difficulty inserting the awl; difficulty putting in the guidewire; Wrong entry point; difficulty finding proximal blade insertion and application; difficulty with distal locking screw determination and insertion
  Any technical difficulty will be described in detail to ascertain the nature and cause of the difficulty (technique dependent vs implant dependent).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meinberg EG, Agel J, Roberts CS, Karam MD, Kellam JF. Fracture and Dislocation Classification Compendium-2018. J Orthop Trauma. 2018 Jan;32 Suppl 1:S1-S170. doi: 10.1097/BOT.0000000000001063. No abstract available. PMID 29256945
- [Background] Chang SM, Zhang YQ, Ma Z, Li Q, Dargel J, Eysel P. Fracture reduction with positive medial cortical support: a key element in stability reconstruction for the unstable pertrochanteric hip fractures. Arch Orthop Trauma Surg. 2015 Jun;135(6):811-8. doi: 10.1007/s00402-015-2206-x. Epub 2015 Apr 4. PMID 25840887
- [Background] Palm H, Jacobsen S, Sonne-Holm S, Gebuhr P; Hip Fracture Study Group. Integrity of the lateral femoral wall in intertrochanteric hip fractures: an important predictor of a reoperation. J Bone Joint Surg Am. 2007 Mar;89(3):470-5. doi: 10.2106/JBJS.F.00679. PMID 17332094
- [Background] Sharma G, kumar G N K, Yadav S, Lakhotia D, Singh R, Gamanagatti S, Sharma V. Pertrochanteric fractures (AO/OTA 31-A1 and A2) not amenable to closed reduction: causes of irreducibility. Injury. 2014 Dec;45(12):1950-7. doi: 10.1016/j.injury.2014.10.007. PMID 25458060
- [Background] Jones HW, Johnston P, Parker M. Are short femoral nails superior to the sliding hip screw? A meta-analysis of 24 studies involving 3,279 fractures. Int Orthop. 2006 Apr;30(2):69-78. doi: 10.1007/s00264-005-0028-0. Epub 2006 Feb 22. PMID 16496147
- [Background] Johnson B, Stevenson J, Chamma R, Patel A, Rhee SJ, Lever C, Starks I, Roberts PJ. Short-term follow-up of pertrochanteric fractures treated using the proximal femoral locking plate. J Orthop Trauma. 2014 May;28(5):283-7. doi: 10.1097/01.bot.0000435629.86640.6f. PMID 24751607
- [Background] Radaideh AM, Qudah HA, Audat ZA, Jahmani RA, Yousef IR, Saleh AAA. Functional and Radiological Results of Proximal Femoral Nail Antirotation (PFNA) Osteosynthesis in the Treatment of Unstable Pertrochanteric Fractures. J Clin Med. 2018 Apr 12;7(4):78. doi: 10.3390/jcm7040078. PMID 29649099
- [Background] Al-yassari G, Langstaff RJ, Jones JW, Al-Lami M. The AO/ASIF proximal femoral nail (PFN) for the treatment of unstable trochanteric femoral fracture. Injury. 2002 Jun;33(5):395-9. doi: 10.1016/s0020-1383(02)00008-6. PMID 12095718
- [Background] Simmermacher RK, Bosch AM, Van der Werken C. The AO/ASIF-proximal femoral nail (PFN): a new device for the treatment of unstable proximal femoral fractures. Injury. 1999 Jun;30(5):327-32. doi: 10.1016/s0020-1383(99)00091-1. PMID 10505125
- [Background] Gardenbroek TJ, Segers MJ, Simmermacher RK, Hammacher ER. The proximal femur nail antirotation: an identifiable improvement in the treatment of unstable pertrochanteric fractures? J Trauma. 2011 Jul;71(1):169-74. doi: 10.1097/TA.0b013e3182213c6e. PMID 21818023
- [Background] Zhou JQ, Chang SM. Failure of PFNA: helical blade perforation and tip-apex distance. Injury. 2012 Jul;43(7):1227-8. doi: 10.1016/j.injury.2011.10.024. Epub 2011 Nov 12. No abstract available. PMID 22079147